CLINICAL TRIAL: NCT06146946
Title: Safety of Mid and Low Rectal Cancer Surgery Without Dissection of the No.253 Lymph Node, a Prospective, Multicenter, Non-inferior Randomized Controlled Trial
Brief Title: Safety of Mid and Low Rectal Cancer Surgery Without Dissection of the No.253 Lymph Node (S-M-O-O-T-H)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Collaborators: Peking Union Medical College Hospital (Other); China-Japan Friendship Hospital (Other); Chinese PLA General Hospital (Other); Ruijin Hospital (Other); Fudan University (Other); West China Hospital (Other); Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, QIAN LIU, Professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC4278
Record Dates: First submitted 2023-11-18; First posted 2023-11-27 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Rectal Cancer
Keywords: Rectal cancer; Lymph node dissection; No.253 lymph node
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Omitting dissection of the No.253 lymph node (Experimental): Perform surgery based on the principle of Total Mesorectal Excision (TME), without denuding the root of the Inferior Mesenteric Artery (IMA) and without dissection of the No.253 lymph node. Ligation of the IMA is performed at a low position distal to the origin of the left colonic artery.
  Interventions: Procedure: Omitting the dissection of the No.253 lymph node
- Dissection of the No.253 lymph node (Active Comparator): Perform surgery based on the principle of Total Mesorectal Excision (TME). During the procedure, fully expose the root of the Inferior Mesenteric Artery (IMA), thoroughly dissect the No.253 lymph node, and perform a high ligation along the artery at the root of the IMA; or expose the bifurcation of the left colonic artery, ligating the IMA at a low position distal to the origin of the left colonic artery, ensuring the dissection of the No. 253 lymph node while preserving the left colonic artery.
  Interventions: Procedure: Dissection of the No.253 lymph node

INTERVENTIONS:
Procedure: Dissection of the No.253 lymph node — The range of the No.253 lymph node is as follows: medially, it extends from the root of the inferior mesenteric artery to the starting section of the left colonic artery; caudally, from the starting point of the left colonic artery to the intersection with the inferior mesenteric vein; laterally, it is bordered by the outer margin of the inferior mesenteric vein; and cranially, from the horizontal section of the duodenum to the beginning of the jejunum. In the controlled group, the surgery is performed with dissection of the No.253 lymph node.
  Arms: Dissection of the No.253 lymph node
Procedure: Omitting the dissection of the No.253 lymph node — In the experimental group, the surgery is performed without dissection of the No.253 lymph node.
  Arms: Omitting dissection of the No.253 lymph node

SUMMARY:
The goal of this clinical trial is to learn about whether it is safe to omit dissection of the No.253 lymph nodes in mid and low rectal cancer surgery. The main question it aims to answer is that if it is possible to achieve the same long-term survival with and without the dissection of the No.253 lymph node in mid and low rectal cancer surgery. Participants will underwent laparoscopic rectal radical resection with or without the dissection of the No.253 lymph node.

DETAILED DESCRIPTION:
The No.253 lymph node, as the third station in the inferior mesenteric artery lymphatic system, plays a significant role in the lymphatic circulation of the descending colon, sigmoid colon, and rectum. They act as the last barrier for tumor metastasis from the regional to distant areas. However, there is still controversy regarding whether rectal cancer patients universally require dissection of the No.253 lymph node. The rate of metastasis to the No.253 lymph node in rectal cancer patients is extremely low, and dissection may not bring survival benefits. Additionally, postoperative urinary and sexual functions may be impaired due to damage to the sympathetic nerves. However, current prospective randomized controlled trials on the safety of omitting the dissection of the No.253 lymph node have small sample sizes and lack sufficient test power. Further confirmation is needed from large-sample prospective randomized controlled studies. Based on this, the investigator plans to collaborate with Peking Union Medical College Hospital, China-Japan Friendship Hospital, Chinese People's Liberation Army General Hospital, Shanghai Ruijin Hospital, Fudan Cancer Hospital, and West China Hospital of Sichuan University, totaling eight medical centers, to conduct a prospective randomized controlled study. This study aims to confirm the safety of mid and low rectal surgery without dissection of the No.253 lymph node, providing high-level evidence-based medical evidence for the implementation of this surgical technique.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age between 18-75 years.
2. Colonic biopsy pathology confirms adenocarcinoma.
3. At initial treatment, colonoscopy and imaging diagnose the tumor's lower edge as less than or equal to 7cm from the anus.
4. At initial treatment, imaging diagnoses the tumor T stage as less than or equal to 3.
5. At initial treatment, imaging diagnoses no enlarged lymph nodes at the root of the inferior mesenteric artery.
6. At initial treatment, imaging diagnoses the number of mesenteric metastatic lymph nodes as less than or equal to three.
7. Strong willingness for surgery and signed informed consent.

Exclusion Criteria:

1. Previous history of malignant colorectal tumors.
2. Colonic biopsy pathology reveals mucinous adenocarcinoma or signet ring cell carcinoma.
3. Imaging diagnosis of distant metastasis.
4. Patients who have undergone multiple abdominal-pelvic surgeries or have extensive abdominal adhesions.
5. Patients with complications such as intestinal obstruction, intestinal perforation, or intestinal bleeding requiring emergency surgery.
6. Extensive lesions not amenable to R0 resection.
7. Diagnosed with other malignancies within the past five years.
8. ASA (American Society of Anesthesiologists) classification ≥ IV and/or ECOG (Eastern Cooperative Oncology Group) performance status score ≥ 2.
9. Patients with severe liver, kidney, cardiac, pulmonary, coagulation dysfunctions, or serious underlying diseases that cannot tolerate surgery.
10. History of severe mental illness.
11. Pregnant or breastfeeding women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1384 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
3-year disease free survival rate | 3 years after surgery
  Disease free survival refers to the length of time after primary treatment during which a patient survives without any signs or symptoms of the cancer.

SECONDARY OUTCOMES:
Number of harvested lymph nodes | About 10 days after surgery
  Total number of lymph nodes dissected in the pathology report
Incidence of postoperative complications | 30 days after surgery
  The proportion of short-term complications occurring within 30 days post-surgery
Intraoperative blood loss | Intraoperative
  Total blood loss during the surgery
Operative duration | Intraoperative
  total time spent performing a surgical procedure. This time is typically measured from the moment the surgery begins (marked by the initial incision) to its conclusion (marked by the closure of the surgical wound)
Postoperative urination and sexual function | 1 year after surgery
  Three months, six months, and one year postoperatively, evaluate patients' urinary and sexual functions using scales.
3-year local recurrence rate | 3 years after surgery
  Local recurrence refers to the return of cancer in the same area where it originally developed, typically after treatment has been completed.
3-year overall survival rate | 3 years after surgery
  Overall survival refers to the length of time from the primary treatment that patients are still alive.

CONTACTS AND LOCATIONS:
Overall Officials: Qian Liu, Principal Investigator — Cancer Hospital Chinese Academy of Medical Science
Locations (8):
- China (8):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijng
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Chaoyang District
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - West China Hospital Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No